CLINICAL TRIAL: NCT07051590
Title: Evaluation of the Time Required for Clinical Adaptation of Partial Dentures Based on Additive and Subtractive Manufacturing: A Randomized Controlled Clinical Study
Brief Title: Adjustment Period for Partial Crowns
Acronym: Adjustment per
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceren Sire (Other)
Responsible Party: Sponsor-Investigator, Ceren Sire, research assistant, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: restorative dentistry
Record Dates: First submitted 2025-06-03; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Deep Caries Lesion of Pemanent Teeth
Keywords: 3D; occlusense; partial crown; cad/cam

STUDY DESIGN:
Intervention Model Description: The subject of this study is to compare the occlusal closure performance of onlay restorations produced from CAD-CAM blocks with onlay restorations produced using 3D printer technology. The Occlusense device has the capacity to measure occlusal contact points and force distribution through digital pressure sensors, providing accurate data in clinical research.
  This study is a randomized clinical trial conducted using a split-mouth design. Onlay restorations produced using different manufacturing methods will be applied to two teeth of the same patient, and the occlusal closures of both restorations will
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- additive (Experimental): manufactured with 3D
  Interventions: Device: 3D printer
- subtractive (Experimental): manufactured with CAD/CAM
  Interventions: Device: cad cam

INTERVENTIONS:
Device: cad cam — Occlusion assessment in CAD CAM restorations
  Arms: subtractive
Device: 3D printer — Crowns produced with 3D technology
  Arms: additive

SUMMARY:
The aim of this study is to compare the occlusal accuracy of CAD/CAM milled and 3D printed crowns guided by an occlusal device, starting from the same digital CAD design.

DETAILED DESCRIPTION:
The subject of this study is to compare the occlusal closure performance of onlay restorations produced from CAD-CAM blocks and onlay restorations produced using 3D printer technology. The Occlusense device has the capacity to measure occlusal contact points and force distribution through digital pressure sensors, providing accurate data in clinical research.

This study is a randomized clinical trial conducted using a split-mouth design. Onlay restorations produced using different manufacturing methods will be applied to two teeth of the same patient, and the occlusal closures of both restorations will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Devitalized and vital teeth with tubercle loss
* ASA I

Exclusion Criteria:

* Teeth with periapical lesions
* Temporomandibular joint disorder or bruxism
* Periodontal disease
* Symptomatic vital teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
crown adjustment times | 1-6 month
  Using the occlusal relationships recorded with the occlusense recorder prior to the restoration preparation as a guide, the occlusal contacts will be adjusted at maximum intercuspation (ICM) and during protrusive and lateral excursive movements. The duration of these adjustments will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: zeliha g bek kürklü, doçent, Study Director — çukurova üniversitesi diş hekimliği restoratif diş tedavisi; Doç. Dr. Dt, Study Director — çukurova üniversitesi diş hekimliği restoratif diş tedavisi
Locations (1):
- Çukurova Üniversitesi, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee WS, Lee DH, Lee KB. Evaluation of internal fit of interim crown fabricated with CAD/CAM milling and 3D printing system. J Adv Prosthodont. 2017 Aug;9(4):265-270. doi: 10.4047/jap.2017.9.4.265. Epub 2017 Aug 16. PMID 28874993